CLINICAL TRIAL: NCT04713501
Title: Program for Alleviating and Resolving Trauma and Stress Study (Stage 1 Pilot)
Brief Title: Program for Alleviating and Resolving Trauma and Stress 1
Acronym: PARTS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Foundation for Self Leadership (Other)
Responsible Party: Principal Investigator, Zev Schuman Olivier, Assistant Professor, Psychiatry, Cambridge Health Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1158/09/20
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: PARTS is a live-online group program intended to alleviate and resolve symptoms of stress and PTSD for patients in a community health care system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PARTS (Experimental): The PARTS Program is a 16-week group intervention model, with 8 individual clinical sessions on a biweekly basis, developed to resolve and alleviate trauma and stress for individuals diagnosed with PTSD.
  Interventions: Behavioral: PARTS Program

INTERVENTIONS:
Behavioral: PARTS Program — The PARTS Program is a 16-week group intervention model, with 8 individual clinical sessions on a biweekly basis, developed to resolve and alleviate trauma and stress for individuals diagnosed with PTSD.

SUMMARY:
This single-arm pilot study (Phase 1) will test the preliminary efficacy of a virtually delivered, live-online 16-week group model of Internal Family Systems (IFS) for individuals with PTSD, called the PARTS program, on PTSD symptoms measured by Clinician-Administered PTSD Scale (CAPS-5). In addition, feasibility, acceptability, and effects on self-report PTSD and disturbances of self-organization (DSO) will be secondary outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a single-arm pilot study to test the preliminary efficacy of a virtually delivered, live-online 16-week group model of Internal Family Systems (IFS) for individuals with PTSD, called the PARTS program, on PTSD symptoms measured by Clinician-Administered PTSD Scale (CAPS-5).

Secondary outcomes include feasibility and acceptability of the PARTS program measured by a Credibility/Expectancy Questionnaire (CEQ) and Treatment Satisfaction Questionnaire. Secondary clinical outcomes include the effects of the PARTS program on self-report PTSD and disturbances of self-organization (DSO). Exploratory aims of the study are to investigate the effects on emotion regulation (DERS), self-trauma fusion (iPRISM-trauma), disassociation (MDI), depression (CAT-DI), self-compassion (SCS-SF), perceived stress (PSS), mindfulness (TMS), and interception (MAIA-2). Additional exploratory outcomes include changes in outcome variables among PTSD subjects with baseline DSO and those without DSO as defined by the International Trauma Questionnaire (ITQ).

ELIGIBILITY:
Inclusion Criteria

To qualify for inclusion in this study, a prospective participant must:

1. Be 18-70 years of age for the duration of the study;
2. Able to bill insurance for group psychotherapy and individual psychotherapy at CHA;
3. Be a current patient of CHA primary care, behavioral health care or CHA MindWell;
4. Have a current diagnosis of PTSD OR a CAT-MH PTSD measure P-CAT>58;
5. Have sufficient English fluency and literacy skills to understand the consent process, procedures and questionnaires and have the ability to provide written informed consent;
6. Have access to the internet and an electronic device with adequate data capacity; to complete questionnaires online and attend online videoconference groups;
7. Must be available and willing to attend the scheduled online group sessions for 16 weeks; and
8. Must be available and willing to complete the online computerized assessments and phone interviews.

Exclusion Criteria

Any and all of the following criteria will exclude a prospective participant from the study:

1. Inability to complete an informed consent assessment AND/OR inability to complete baseline study assessment procedures (due to cognitive deficit, non- proficiency in English literacy, or for any other reason);
2. Current participation in another experimental research study;
3. Expected medical hospitalization in the next six months from enrollment period;
4. Expected incarceration in the next six months from enrollment period;
5. Individuals who are pregnant with a due date within 26 weeks after study consent;
6. Insufficient level of severity of PTSD symptoms: PTSD score of less than 33 on the PTSD Checklist for DSM-V (PCL-5) at screening visit;
7. Inability to participate safely in the study intervention and without disrupting the group (in the opinion of principal investigator OR meeting any of the following criteria):

   * Past year history of a psychotic disorder or clinician confirmed active psychosis (Severe level of psychosis on PSY-S-CAT > 60 will trigger the requirement of a clinical assessment prior to participation in the program)
   * Bipolar I disorder history or severe level of mania on CAT-M/HM (>70)
   * Acute suicidality or self-injurious behavior
   * Severe depression, indicated by CAT-DI PHQ-9 equivalency score >20
   * Acute homicidality with plan and/or intent;
   * Hospitalization for suicide attempt or self-harm within three months of the enrollment period;
   * Severe Borderline Personality Disorder or other severe personality disorder that may lead to disruptions within the group; and/or
   * Moderate or severe Substance Use Disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline CAPS-5 at 16 Weeks | Week 16
  The primary aim of this study is to examine the preliminary efficacy of a live-online version of the PARTS program on PTSD symptoms measured by reduction in CAPS-5 over 24 weeks. The CAPS-5 is a 30-item questionnaire administered by a trained interviewer and is considered the "gold standard" assessment for PTSD diagnosis and symptoms as defined by the DSM-5. This measure also assesses the duration of symptoms, impact of symptoms on aspects of the participant's life, and if the participant meets criteria for the dissociative subtype of PTSD.

SECONDARY OUTCOMES:
Retention | Week 16
  A secondary aim is to evaluate feasibility by demonstrating at least 50% of participants are retained in the program at 16 weeks..
Acceptability as assessed by Satisfaction Survey | Week 16
  Participants will complete a satisfaction survey and rate their likeliness to recommend the program to a friend, on a five point Likert-type scale. An average greater than 3 out of 5 represents acceptability.
Change from Baseline Self-reported PTSD symptoms (PCL-5) at 16 Weeks | Week 16
  Participants will be sent a link to complete the PTSD Checklist for DSM-5 (PCL-5), which is a self-report measure with 20 items, which is designed to measure PTSD symptom severity over the past month as measured by the DSM-5, in combination with additional diagnostic tools.
Change from Baseline Self-reported PTSD symptoms (CAT-PTSD) at 16 Weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome refers to the CAT-PTSD severity score
Change from Baseline Disturbances of Self Organization -- International Trauma Questionnaire (ITQ-DSO-9) at 16 Weeks | Week 16
  The International Trauma Questionnaire (ITQ) is the first instrument designed to capture the ICD-11 PTSD and Complex PTSD (CPTSD) diagnoses. The last 6 items measure DSO symptoms characteristic of ICD-11 CPTSD. Each set of items have 3 severity of impact on functioning questions. The ITQ-DSO-9 includes just the 6 DSO items with 3 severity questions. The ITQ-DSO-9 will be used monthly for self-report of changes in DSO symptoms.

OTHER OUTCOMES:
Change from Baseline Difficulties in Emotion Regulation (DERS) Scale at 16 Weeks | Week 16
  The DERS is a 36-item self-report scale designed to assess emotional dysregulation. The scale assess 6 aspects of emotional dysregulation: non-acceptance of emotional responses ("When I'm upset, I become embarrassed for feeling that way"), difficulties engaging in goal directed behavior ("When I'm upset, I have difficulty thinking about anything else"), impulse control difficulties ("When I'm upset, I lose control over my behaviors"), lack of emotional awareness ("When I'm upset, I take time to figure out what I'm really feeling (reverse-scored)", limited access to emotion regulation strategies ("When I'm upset, it takes me a long time to feel better"), and lack of emotional clarity ("I have no idea how I am feeling").
Change from Baseline Pictorial Representation of Illness and Self Measure (PRISM) --Trauma at 16 Weeks | Week 16
  The Pictorial Representation of Illness and Self Measure (PRISM) is a visual method to assess the global burden of illness, measuring the participant's "self-trauma fusion". Using the iPrism Lite ipad app, the user places a disk representing the illness in relation to a disk representing the self.
Change from Baseline Multiscale Dissociation Inventory (MDI) at 16 Weeks | Week 16
  The MDI is a 30-item self-report inventory measuring frequency of dissociative symptoms (e.g., depersonalization, derealization, emotional constriction, identity dissociation, etc.)
Change from Baseline Depression (CAT-DI) at 16 Weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assess depression severity with the CAT-DI.
Change from Baseline Self-Compassion Scale (SCS-SF) at 16 Weeks | Week 16
  The SCS-SF is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. This scale evaluates 6 different aspects of self-compassion: Self-Kindness (e.g., ''I try to be understanding and patient toward those aspects of my personality I don't like''), Self-Judgment (e.g., ''I'm disapproving and judgmental about my own flaws and inadequacies''), Common Humanity (e.g., ''I try to see my failings as part of the human condition''), Isolation (e.g., ''When I feel inadequate in some way, I try to remind myself that feelings of inadequacy are shared by most people"), Mindfulness (e.g., ''When something painful happens I try to take a balanced view of the situation''), and Over-Identification (e.g., ''When I'm feeling down I tend to obsess and fixate on everything that's wrong.''). The scale is scored on a 5-point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored.
Change from Baseline Perceived Stress Scale (PSS-4) at 16 Weeks | Week 16
  The PSS-4 uses 4 items to measure the degree to which situations in life are stressful, evaluating how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5-point Likert scale from 0 (Never) to 4 (Very often).
Change from Baseline Toronto Mindfulness Scale (TMS) at 16 Weeks | Week 16
  The TMS is a 13-item scale evaluating mindfulness factors of curiosity and decentering.
Change from Baseline Multidimensional Assessment of Interoceptive Awareness (MAIA-2) at 16 Weeks | Week 16
  The MAIA-2 is a 37-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness (e.g., body trusting).

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Eisen SV, Schultz MR, Ni P, Haley SM, Smith EG, Spiro A, Osei-Bonsu PE, Nordberg S, Jette AM. Development and Validation of a Computerized-Adaptive Test for PTSD (P-CAT). Psychiatr Serv. 2016 Oct 1;67(10):1116-1123. doi: 10.1176/appi.ps.201500382. Epub 2016 Jun 1. PMID 27247175
- [Background] Wittmann L, Schnyder U, Buchi S. PRISM (Pictorial Representation of Illness and Self Measure): a new method for the assessment of suffering after trauma. J Trauma Stress. 2012 Feb;25(1):94-7. doi: 10.1002/jts.20710. Epub 2012 Jan 25. PMID 22278709
- [Background] Briere J, Weathers FW, Runtz M. Is dissociation a multidimensional construct? Data from the Multiscale Dissociation Inventory. J Trauma Stress. 2005 Jun;18(3):221-31. doi: 10.1002/jts.20024. PMID 16281216
- [Background] Achtyes ED, Halstead S, Smart L, Moore T, Frank E, Kupfer DJ, Gibbons R. Validation of Computerized Adaptive Testing in an Outpatient Nonacademic Setting: The VOCATIONS Trial. Psychiatr Serv. 2015 Oct;66(10):1091-6. doi: 10.1176/appi.ps.201400390. Epub 2015 Jun 1. PMID 26030317
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Mitchell AM, Crane PA, Kim Y. Perceived stress in survivors of suicide: psychometric properties of the Perceived Stress Scale. Res Nurs Health. 2008 Dec;31(6):576-85. doi: 10.1002/nur.20284. PMID 18449942
- [Background] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Gratz, K.L., Roemer, L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26, 41-54 (2004). https://doi.org/10.1023/B:JOBA.0000007455.08539.94